CLINICAL TRIAL: NCT02836574
Title: A Phase 2 Prospective, Randomized, Double-Arm, Deferred Treatment, Open Label, Repeat Dose, Safety and Efficacy Study of Renal Autologous Cell Therapy (REACT) in Subjects With Type 2 Diabetes and Chronic Kidney Disease
Brief Title: A Study of Renal Autologous Cell Therapy (REACT) in Type 2 Diabetics With Chronic Kidney Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prokidney (Industry)
Collaborators: CTI Clinical Trial and Consulting Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RMCL-002
Record Dates: First submitted 2016-06-22; First posted 2016-07-19 (Estimated); Last update posted 2025-08-24 (Actual); Status verified 2024-10

CONDITIONS: Type 2 Diabetes Mellitus; Chronic Kidney Disease
Keywords: Rilparencel
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Treatment (Experimental): Renal Autologous Cell Therapy (REACT) immediate treatment - Patients who are randomized to receive their first treatment of 2 injections of REACT as soon as REACT product is made available.
  Interventions: Biological: Renal Autologous Cell Therapy (REACT); Procedure: Renal Biopsy
- Deferred Treatment (Active Comparator): Renal Autologous Cell Therapy (REACT) delayed treatment - Patients who are randomized to receive standard of care treatment for the first 12 months after REACT product is made available before receiving 2 injections of REACT.
  Interventions: Biological: Renal Autologous Cell Therapy (REACT); Procedure: Renal Biopsy

INTERVENTIONS:
Biological: Renal Autologous Cell Therapy (REACT) — Autologous selected renal cells (SRC).
  Other Names: Rilparencel
Procedure: Renal Biopsy — a procedure in which a small sample of kidney tissue is removed
  Other Names: Kidney Biopsy

SUMMARY:
To assess the safety and efficacy of up to two REACT injections given 6 months (+4 weeks) apart and delivered into the biopsied kidney using a percutaneous approach in participants with Type 2 Diabetes Mellitus (T2DM) and Chronic Kidney Disease (CKD).

DETAILED DESCRIPTION:
Study Part 1: Multi-center, prospective, open-label, randomized, double-arm, deferred treatment study whereby eligible subjects will be randomized 1:1 after kidney biopsy to receive up to 2 injections of REACT (made from expanded autologous selected renal cells) into the biopsied kidney beginning as soon as REACT can be prepared, or the same series of up to 2 injections given 6 months (+4 weeks) apart beginning 12 months after renal biopsy. Subjects will be followed through 23 months after the last injection.

Study Part 2: An open-label extension study in which eligible subjects will be followed for an additional 36 months of long-term follow-up. Subjects will be able to roll from Study Part 2 into a Long Term Follow-Up Master protocol for up to 5 years

ELIGIBILITY:
Inclusion Criteria for Study Part 1:

1. The subject is male or female, 30 to 80 years of age on the date of informed consent.
2. The subject has an established diagnosis of Type 2 Diabetes Mellitus.
3. The subject has an established diagnosis of diabetic nephropathy as the underlying cause of renal disease.
4. The subject has an established diagnosis of Chronic Kidney Disease not requiring renal dialysis, defined as having an Estimated Glomerular Filtration Rate (eGFR) between 20 and 50 mL/min/1.73m².
5. The subject has blood pressure less than 150/90 at the Screening Visit.
6. The subject has stable blood pressure and is maintained on a stable anti-hypertensive medication regimen.
7. A minimum of 2 measurements of Estimated Glomerular Filtration Rate (eGFR) or serum creatine ratio (sCr) should be obtained at least 3 months apart prior to the Screening Visit or within the previous 18 months to define the rate of progression of Chronic Kidney Disease (CKD).

Exclusion Criteria for Study Part 1:

1. The subject has a history of type 1 diabetes mellitus.
2. The subject has a history of renal transplantation.
3. The subject has a serum Hemoglobin A1c (HbA1c) level greater than 10% at the Screening Visit.
4. The subject has uncontrolled diabetes (defined as metabolically unstable by the Investigator).
5. The subject has hemoglobin levels less than 9 g/dL prior to each Renal Autologous Cell Therapy (REACT) injection.

Inclusion Criteria for Study Part 2:

1. The subject is willing and able to provide signed informed consent.
2. The subject was enrolled into Part 1 of the study and received at least one Renal Autologous Cell Therapy (REACT) injection.

Exclusion Criteria for Study Part 2:

1. The subject is currently receiving renal dialysis.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2023-12 (Actual); Study Completion 2023-12 (Actual)

PRIMARY OUTCOMES:
Change in Renal Function | Through 24 months following last REACT injection for active arm and at least 12 months following last REACT injection for the deferred arm
  Serial measurements of estimated glomerular filtration rate (eGFR) obtained pre-randomization and at three-month intervals through 24 months after the last REACT injection in the active treatment group and at least 12 months post last REACT injection in the deferred treatment group.

SECONDARY OUTCOMES:
Treatment emergent adverse events | Through 24 months following last REACT injection for the active arm and at least 12 months following the last REACT injection for the deferred arm
  Treatment emergent adverse events, serial safety laboratory results

CONTACTS AND LOCATIONS:
Overall Officials: Brian Johnston, Study Director — CTI
Locations (16):
- United States (16):
  - University of Arizona, Tucson, Arizona
  - Kidney Associates of Colorado, Denver, Colorado
  - Yale Univeristy, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - Boise Kidney and Hypertension Institute, Meridian, Idaho
  - University of Chicago Medical Center, Chicago, Illinois
  - University of Louisville, Louisville, Kentucky
  - Renal Associates of Baton Rouge, Baton Rouge, Louisiana
  - University of Michigan, Ann Arbor, Michigan
  - Paragon Health, Kalamazoo, Michigan
  - Nephrology & Hypertension Associates, Tupelo, Mississippi
  - Mt. Sinai Hospital, New York, New York
  - University of North Carolina- Chapel Hill, Chapel Hill, North Carolina
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - University of Wisconsin-Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stavas J, Gerber D, Coca SG, Silva AL, Johns A, Jain D, Bertram T, Diaz-Gonzalez de Ferris M, Bakris G. Novel Renal Autologous Cell Therapy for Type 2 Diabetes Mellitus Chronic Diabetic Kidney Disease: Clinical Trial Design. Am J Nephrol. 2022;53(1):50-58. doi: 10.1159/000520231. Epub 2022 Jan 14. PMID 35034024